CLINICAL TRIAL: NCT04732949
Title: A Randomised, Double-blind, Placebo-controlled, Phase III Trial to Determine the Efficacy and Safety of Inhaled SNG001 for the Treatment of Patients Hospitalised Due to Moderate COVID-19
Brief Title: Study to Assess Efficacy and Safety of Inhaled Interferon-β Therapy for COVID-19
Acronym: SPRINTER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Synairgen Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SG018; 2020-004743-83 (EudraCT Number)
Record Dates: First submitted 2021-01-28; First posted 2021-02-01 (Actual); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2021-01

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2; COVID-19
Keywords: Coronavirus disease-2019 (COVID-19); Interferon beta
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study will be patient and investigator-blinded with regard to SNG001 or placebo but not the dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SNG001 (Active Comparator): SNG001 via inhalation using Ultra device, once a day for 14 days
  Interventions: Drug: SNG001
- Placebo (Placebo Comparator): Placebo via inhalation using Ultra device, once a day for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SNG001 — SNG001 nebuliser solution, 2 syringes each containing 0.65 mL once a day
  Arms: SNG001
Drug: Placebo — Placebo nebuliser solution, 2 syringes each containing 0.65 mL solution containing excipients of the SNG001 solution
  Arms: Placebo

SUMMARY:
The purpose of this Phase III study is to confirm that SNG001 can accelerate the recovery of hospitalised patients receiving oxygen with confirmed Severe Acute Respiratory Syndrome coronavirus 2 (SARS-CoV-2). Safety and other efficacy endpoints will also be assessed.

DETAILED DESCRIPTION:
Eligible patients with SARS-CoV-2 infection confirmed by a positive virus test and who are hospitalised due to COVID-19 and require oxygen therapy, will be randomised in a 1:1 ratio to receive SNG001 two syringes or placebo two syringes. SNG001 or placebo will be administered via the Ultra nebuliser. Patients will receive a dose of SNG001 or placebo once a day for 14 days and will be followed up for up to 90 days after the first dose of study medication. Study data will be collected from patients daily, as per the study schedule.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital due to the severity of their COVID-19
* Positive virus test for SARS-CoV-2 using a validated molecular assay or antigen assay. Patients who had a positive virus test for SARS-CoV-2 prior to hospitalisation will be randomised no later than 48 hours after hospital admission. If the virus test is performed more than 96 hours prior to hospitalisation, the test will have to be repeated in the hospital prior to randomisation. Only patients whose repeated virus test is positive will be randomised, no later than 48 hours after confirmation of SARS-CoV-2 infection. Patients who had their first positive virus test for SARS-CoV-2 after hospitalisation will be randomised no later than 48 hours after confirmation of SARS-CoV-2 infection
* Require oxygen therapy via nasal prongs or mask (WHO OSCI score of 4)
* Provided informed consent
* Female patients must be ≥1 year post-menopausal, surgically sterile, or using a protocol defined highly effective method of contraception
* Women of child bearing potential should have been stable on their chosen method of birth control for a minimum of 3 months before entering the trial and should continue with birth control for 1 month after the last dose of inhaled interferon-β (IFN-β1a)/matching placebo. In addition to the highly effective method of contraception (except for the practice of total sexual abstinence), a condom (in United Kingdom with spermicides) should be used by the male partner for sexual intercourse from randomisation (Visit 2) and for 1 month after the last dose of inhaled IFN-β1a/matching placebo to prevent pregnancy
* Women not of childbearing potential are defined as women who are either permanently sterilised (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months prior to the planned date of randomisation without an alternative medical cause. The following age specific requirements apply: women <50 years old will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and if follicle stimulating hormone (FSH) levels are in the postmenopausal range; women ≥50 years old will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatment. If, in the setting of the pandemic, the use of an acceptable birth control method is not possible, the decision to enrol a woman of childbearing potential should be based on the benefit-risk for the patient, which should be discussed with the patient at the time of the informed consent.

Exclusion Criteria:

* Evidence of ongoing SARS-CoV-2 infection for more than 3 weeks, confirmed by a validated molecular assay or validated antigen assay
* Non-invasive ventilation continuous positive airway pressure/bilevel positive airway pressure (CPAP/BiPAP) or high-flow nasal oxygen therapy (WHO OSCI score of 5)
* Endotracheal intubation and invasive mechanical ventilation (WHO OSCI score of ≥6) or admission to intensive care
* Previous SARS-CoV-2 infection confirmed by a validated molecular assay or validated antigen assay
* Any condition, including findings in the patients' medical history or in the pre-randomisation study assessments that in the opinion of the Investigator, constitute a risk or a contraindication for the participation of the patient into the study or that could interfere with the study objectives, conduct or evaluation
* Participation in previous clinical trials of SNG001
* Current or previous participation in another clinical trial where the patient has received a dose of an Investigational Medicinal Product containing small molecules within 30 days or 5 half-lives (whichever is longer) prior to entry into this study or containing biologicals within 3 months prior to entry into this study
* Inability to use a nebuliser with a mouthpiece
* Inability to comply with the requirements for storage conditions of study medication in the home setting
* History of hypersensitivity to natural or recombinant IFN-β or to any of the excipients in the drug preparation
* Females who are breast-feeding, lactating, pregnant or intending to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Tom Wilkinson, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (112):
- United States (6):
  - The University of Arizona Medi, Tucson, Arizona
  - Professional Health Care of Pi, St. Petersburg, Florida
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Icahn School of Medicine at Mo, New York, New York
  - PharmaTex Research, LLC, Amarillo, Texas
- Argentina (3):
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, Ciudad Autónoma de Buenos Air, Buenos Aires
  - Hospital Universitario Austral, Buenos Aires
  - Hospital Papa Francisco - Hosp, Salta
- Belgium (5):
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - Centre Hospitalier Universitai, Brussels
  - UZ Brussel - Campus Jette - In, Brussels
  - CHR de la Citadelle - Site Cit, Liège
  - CHU de Liège - Domaine Univers, Liège
- Brazil (6):
  - Instituto Mederi de Pesquisa e Saúde, Passo Fundo, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Clínica SUPERA, Chapecó, Santa Catarina
  - Sociedade Literaria e Caritativa Santo Agostinho, Criciúma, Santa Catarina
  - Instituto de Pesquisa Clínica, Campinas, São Paulo
  - Fundacao Faculdade Regional de, São José do Rio Preto, São Paulo
- Colombia (3):
  - Clinica de la Mujer, Bogotá, Cundinamarca
  - FOSCAL, Bucaramanga, Santander Department
  - Clinica de la Costa, Barranquilla
- France (6):
  - CHU De Nantes - Infectious Dis, Nantes, Loire-Atlantique
  - CHU d'Angers, Angers, Pays de la Loire Region
  - CHU de Grenoble - Hôpital Albe, La Tronche
  - CHU Saint Antoine - Infectious, Paris
  - Hôpital Européen Georges-Pompi, Paris
  - Hopital Bichat - Infectious Di, Paris
- Germany (3):
  - RoMed Medical Center Rosenheim, Rosenheim, Bavaria
  - Universitätsklinikum Mannheim, Mannheim
  - Krankenhaus Bethanien gGmbH, Solingen
- India (13):
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Unity Hospital, Surat, Gujarat
  - Rhythm Heart Institute, Vadodara, Gujarat
  - Bangalore Medical College and Research Institute, Bangalore, Karnataka
  - MS Ramaiah Medical College and Hospital, Bangalore, Karnataka
  - Oriion Citicare Super Speciality Hospital - Intern, Aurangabad, Maharashtra
  - Fortis Hospital Mulund - Inter, Mumbai, Maharashtra
  - Government Medical College Nag, Nagpur, Maharashtra
  - Suyog Hospital, Nashik, Maharashtra
  - Vishwa Raj Hospital, Pune, Maharashtra
  - Acharya Vinoba Bhave Rural Hos, Wardha, Maharashtra
  - Post Graduate Institute of Medical Education & Research, Chandigarh, Chandigarh, Punjab
  - Saveetha Medical College & Hospital, Chennai
- Israel (6):
  - Assuta Ashdod University Hospi, Ashdod, Southern District
  - Rambam Health Care Campus, Haifa
  - Ziv Medical Center, Safed
  - Sourasky Tel Aviv Medical Cent, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (9):
  - Azienda Socio Sanitaria Territ, Monza, Lombardy
  - Azienda Ospedaliera Nazionale, Alessandria
  - PO A.Manzoni di Lecco, ASST Le, Lecco
  - Ospedale Luigi Sacco, AO-PU, Milan
  - Azienda Ospedaliera Ospedale N, Milan
  - AOU Federico II - Malattie Inf, Napoli
  - IRCCS Policlinico San Matteo, Pavia
  - AOU Pisana, Pisa
  - Città della Salute e della Scienza, Torino
- Mexico (5):
  - Fundación Santos y de la Garza Evia, I.B.P, Monterrey, Nuevo León
  - Hospital General de Culiacan D, Culiacán, Sinaloa
  - EME RED Hospitalaria - COVID-1, Mérida, Yucatán
  - Hospital General Regional O´Hu, Mérida, Yucatán
  - Clínica Sociedad Española de Beneficencia, Veracruz
- Netherlands (3):
  - Ziekenhuis St Jansdal, Harderwijk, Gelderland
  - Gelre Ziekenhuis Zutphen, Zutphen, Gelderland
  - Isala Klinieken, Zwolle, Overijssel
- Portugal (5):
  - Hospital Garcia da Orta, E.P.E, Almada, Lisbon District
  - C.H. de Vila Nova de Gaia/Espi, Vila Nova de Gaia, Porto District
  - Hospital de Braga, Braga
  - Hospital da Senhora de Oliveir, Guimarães
  - Centro Hospitalar de Entre Dou, Rodrigues
- Romania (4):
  - Sp. Clinic Boli Infectioase si, Timișoara, Timiș County
  - Spitalul Universitar de Urgent, Bucharest
  - Sp. Cl. de Boli Infectioase si, Bucharest
  - Spitalul Clinic de Boli Infect, Craiova
- Serbia (5):
  - Clinical Center Nis, Niš, Nišavski Okrug
  - Clinical Center of Vojvodina, Novi Sad, Vojvodina
  - University Clinical Center of Serbia, Belgrade
  - The Institute for Pulmonary Di, Kamenitz
  - Clinical Center Kragujevac, Cl, Kragujevac
- Spain (10):
  - CHU A Coruña, Madrid, A Coruña
  - Hospital Universitario Son Esp, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Mutua d, Terrassa, Barcelona
  - Hospital Universitario de Puer, Puerto Real, Cádiz
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Infanta, Madrid
  - Hospital Universitario Ramón y, Madrid
  - H.Clinico San Carlos, Madrid
  - Hospital Universitario de Sala, Salamanca
  - H U Nuesta Señora de Valme - I, Seville
- United Kingdom (20):
  - Wexham Park Hospital, Slough, Bracknell Forest
  - Hull Royal Infirmary, Hull, North Humberside, East Riding Of Yorkshire
  - Newcastle University - Institute of Cellular Medicine (ICM), Newcastle, England
  - Southampton General Hospital, Southampton, Hampshire
  - Churchill Hospital, Headington, Oxfordshire
  - Frimley Park Hospital, Frimley, Surrey
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - The Royal Bournemouth & Christ, Bournemouth
  - University Hospital of North D, Durham
  - Royal Devon & Exeter Hospital, Exeter
  - Glasgow Royal Infirmary, Glasgow
  - Glenfield Hospital, Leicester
  - University Hospital Lewisham, London
  - Guy's Hospital, London
  - North Manchester General Hospi, Manchester
  - The James Cook University Hosp, Middlesbrough
  - Nottingham University Hospital, Nottingham
  - Plymouth Hospitals NHS Trust, Plymouth
  - Morriston Hospital Swansea NHS, Swansea
  - University Hospital of Wales, Swansea

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 112 centers which included 623 patients across 17 countries. The trial began on 12 January 2021 (first patient consented) and was completed on 10 Feb 2022.
Pre-assignment Details: The pre-treatment assessments were performed on Day 0 prior to the first dose preferably. All the study assessments were performed as per the schedule of assessments.
Groups:
- SNG001: Patients received SNG001 via inhalation using nebuliser, once a day for 14 days
- Placebo: Patients received Placebo via inhalation using nebuliser, once a day for 14 days
Period: Overall Study
Arm/Group | SNG001 | Placebo
Started | 309 | 314
Completed | 233 | 231
Not Completed | 76 | 83
Not completed — Withdrawal by Subject | 23 | 27
Not completed — Protocol Violation | 0 | 1
Not completed — Non-compliance | 0 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Serious adverse event (Fatal) | 16 | 18
Not completed — Serious adverse event (Non fatal) | 2 | 1
Not completed — Non-serious adverse event | 1 | 3
Not completed — Lost to Follow-up | 26 | 27
Not completed — Other | 6 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) analysis population consisted of all randomised patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | SNG001 | Placebo | Total
Number analyzed (Participants) | 309 | 314 | 623
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (15.19) | 53.7 (14.42) | 52.8 (14.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 208 | 411
  Male | 106 | 106 | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 53 | 49 | 102
  Not Hispanic or Latino | 238 | 242 | 480
  Unknown or Not Reported | 18 | 23 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 224 | 215 | 439
  Black | 7 | 6 | 13
  Asian- Chinese | 2 | 2 | 4
  Asian- Other | 40 | 46 | 86
  Arab | 2 | 5 | 7
  American Indian | 5 | 5 | 10
  Other | 10 | 13 | 23
  Unknown | 19 | 22 | 41

OUTCOME MEASURES:

1. Primary Outcome: Time to Hospital Discharge
Description: The time to hospital discharge in patients with moderate COVID-19 after administration of SNG001 compared to placebo was evaluated.
Time Frame: Day 28
Population: The Intent-to-Treat (ITT) analysis population consisted of all randomised patients.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 309 | 314
days | 7.0 [7.0 to 8.0] | 8.0 [7.0 to 9.0]
Statistical Analysis 1: Comparison: SNG001 vs Placebo; Hazard Ratio for time to hospital discharge - SNG001 vs Placebo; Test type: Other; p = 0.509, Cox proportional hazard model; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.89 to 1.27]

2. Primary Outcome: Time to Recovery
Description: Recovery in patients with moderate COVID-19 after administration of SNG001 compared to placebo by time to recovery was evaluated.
Time Frame: Day 28
Population: The ITT analysis population consisted of all randomised patients.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 309 | 314
days | 25.0 [22.0 to NA] — Not calculable due to Insufficient number of participants with events | 25.0 [22.0 to NA] — Not calculable due to Insufficient number of participants with events
Statistical Analysis 1: Comparison: SNG001 vs Placebo; Hazard Ratio for time to OSCI recovery - SNG001 vs Placebo; Test type: Other; p = 0.888, Cox proportional hazard model; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.81 to 1.28]

3. Secondary Outcome: Number of Patients Who Progressed to Severe Disease or Death
Description: The efficacy of SNG001 compared to placebo in patients with moderate COVID-19 by assessing progression to severe disease or death was evaluated. Severe disease was defined by the Ordinal Scale for Clinical Improvement (OSCI) as a score between 5 and 7. Death was defined by an OSCI score of 8.
Time Frame: Until Day 35
Population: The ITT analysis population consisted of all randomised patients. Here, the number of participants analyzed signifies the participants with available data that were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 308 | 312
Participants | 33 | 45
Statistical Analysis 1: Comparison: SNG001 vs Placebo; Odds Ratio for progression to severe disease or death - SNG001 vs Placebo; Test type: Other; p = 0.161, Regression, Logistic; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.44 to 1.15]

4. Secondary Outcome: Number of Patients Who Were Intubated or Who Died
Description: The efficacy of SNG001 compared to placebo in patients with moderate COVID-19 by assessing progression to intubation or death was evaluated. Intubation was defined by the OSCI as a score between 6 and 7. Death was defined by an OSCI score of 8.
Time Frame: Until Day 35
Population: The ITT analysis population consisted of all randomised patients.
Measure: Count of Participants; unit: Participants
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 309 | 314
Participants | 20 | 23
Statistical Analysis 1: Comparison: SNG001 vs Placebo; Odds Ratio for intubation or death - SNG001 vs Placebo; Test type: Other; p = 0.610, Regression, Logistic; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.45 to 1.61]

5. Secondary Outcome: Number of Patients Who Died Within 35 Days of First Dose
Description: Patients who died within 35 days of first dose of study intervention were calculated.
Time Frame: Until Day 35 of first dose
Population: The ITT analysis population consisted of all randomised patients.
Measure: Count of Participants; unit: Participants
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 309 | 314
Participants | 14 | 17
Statistical Analysis 1: Comparison: SNG001 vs Placebo; Odds Ratio for death - SNG001 vs Placebo; Test type: Other; p = 0.544, Regression, Logistic; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.38 to 1.67]

6. Secondary Outcome: Cumulative Number of Patients Who Were Discharged From Hospital
Description: The efficacy of SNG001 compared to placebo in patients with moderate COVID-19 was assessed by hospital discharge on given days.
Time Frame: Days 7, 14, 21 and 28
Population: The ITT analysis population consisted of all randomised patients.
Measure: Count of Participants; unit: Participants
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 309 | 314
Participants
  Day 7 | 154 | 141
  Day 14 | 231 | 223
  Day 21 | 245 | 249
  Day 28 | 249 | 255
Statistical Analysis 1: Comparison: SNG001 vs Placebo; Odds Ratio for hospital discharge (Day 7) - SNG001 vs Placebo; Test type: Other; p = 0.323, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.85 to 1.64]
Statistical Analysis 2: Comparison: SNG001 vs Placebo; Odds Ratio for hospital discharge (Day 14) - SNG001 vs Placebo; Test type: Other; p = 0.406, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.81 to 1.70]
Statistical Analysis 3: Comparison: SNG001 vs Placebo; Odds Ratio for hospital discharge (Day 21) - SNG001 vs Placebo; Test type: Other; p = 0.828, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.64 to 1.43]
Statistical Analysis 4: Comparison: SNG001 vs Placebo; Odds Ratio for hospital discharge (Day 28) - SNG001 vs Placebo; Test type: Other; p = 0.706, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.61 to 1.40]

7. Secondary Outcome: Cumulative Number of Patients With Recovery
Description: The efficacy of SNG001 compared to placebo in patients with moderate COVID-19 by assessing recovery was evaluated. Recovery is defined as no limitation of activities according to the Ordinal Scale of Clinical Improvement (OSCI), with no rebound at subsequent assessments.
Time Frame: Days 7, 14, 21 and 28
Population: The ITT analysis population consisted of all randomised patients.
Measure: Count of Participants; unit: Participants
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 309 | 314
Participants
  Day 7 | 28 | 17
  Day 14 | 75 | 73
  Day 21 | 117 | 118
  Day 28 | 145 | 151
Statistical Analysis 1: Comparison: SNG001 vs Placebo; Odds Ratio for OSCI recovery (Day 7) - SNG001 vs Placebo; Test type: Other; p = 0.101, Regression, Logistic; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.90 to 3.22]
Statistical Analysis 2: Comparison: SNG001 vs Placebo; Odds Ratio for OSCI recovery (Day 14) - SNG001 vs Placebo; Test type: Other; p = 0.942, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.67 to 1.45]
Statistical Analysis 3: Comparison: SNG001 vs Placebo; Odds Ratio for OSCI recovery (Day 21) - SNG001 vs Placebo; Test type: Other; p = 0.824, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.68 to 1.35]
Statistical Analysis 4: Comparison: SNG001 vs Placebo; Odds Ratio for OSCI recovery (Day 28) - SNG001 vs Placebo; Test type: Other; p = 0.613, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.66 to 1.28]

8. Secondary Outcome: Improvement Based on Entire WHO OSCI Score
Description: The efficacy of SNG001 compared to placebo in patients with moderate COVID-19 by assessing improvement across the entire WHO OSCI were evaluated. Improvement in clinical status is based on the 9-point OSCI score. The score ranges from 0 to 8, where lower score of 0 represents no clinical or virological evidence of infection and higher score of 8 represents death.Higher scores indicated worse outcome.
Time Frame: Until Day 35
Measure: Count of Participants; unit: Participants
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 309 | 314
Participants
  Baseline: 0 = No clinical or virological evidence of infection | 0 | 0
  Baseline: 1 = No limitations of activities | 0 | 0
  Baseline: 2 = Limitation of activities | 1 | 0
  Baseline: 3 = Hospitalised - no oxygen therapy | 3 | 8
  Baseline: 4 = Oxygen by mask, or nasal prongs | 304 | 304
  Baseline: 5 = Non-invasive ventilation, or high flow oxygen | 1 | 2
  Baseline: 6 = Intubation and mechanical ventilation | 0 | 0
  Baseline: 7 = Ventilation plus additional organ support | 0 | 0
  Baseline: 8 = Death | 0 | 0
  Baseline: Missing | 0 | 0
  Day 7: 0 = No clinical or virological evidence of infection | 20 | 14
  Day 7: 1 = No limitations of activities | 18 | 12
  Day 7: 2 = Limitation of activities | 115 | 114
  Day 7: 3 = Hospitalised - no oxygen therapy | 42 | 42
  Day 7: 4 = Oxygen by mask, or nasal prongs | 53 | 69
  Day 7: 5 = Non-invasive ventilation, or high flow oxygen | 18 | 26
  Day 7: 6 = Intubation and mechanical ventilation | 2 | 2
  Day 7: 7 = Ventilation plus additional organ support | 3 | 3
  Day 7: 8 = Death | 4 | 0
  Day 7: Missing | 34 | 32
  Day 14: 0 = No clinical or virological evidence of infection | 62 | 57
  Day 14: 1 = No limitations of activities | 24 | 30
  Day 14: 2 = Limitation of activities | 135 | 127
  Day 14: 3 = Hospitalised - no oxygen therapy | 11 | 18
  Day 14: 4 = Oxygen by mask, or nasal prongs | 13 | 15
  Day 14: 5 = Non-invasive ventilation, or high flow oxygen | 2 | 4
  Day 14: 6 = Intubation and mechanical ventilation | 3 | 1
  Day 14: 7 = Ventilation plus additional organ support | 3 | 9
  Day 14: 8 = Death | 9 | 7
  Day 14: Missing | 47 | 46
  Day 21: 0 = No clinical or virological evidence of infection | 89 | 94
  Day 21: 1 = No limitations of activities | 32 | 23
  Day 21: 2 = Limitation of activities | 109 | 114
  Day 21: 3 = Hospitalised - no oxygen therapy | 3 | 4
  Day 21: 4 = Oxygen by mask, or nasal prongs | 7 | 4
  Day 21: 5 = Non-invasive ventilation, or high flow oxygen | 1 | 0
  Day 21: 6 = Intubation and mechanical ventilation | 2 | 1
  Day 21: 7 = Ventilation plus additional organ support | 2 | 8
  Day 21: 8 = Death | 12 | 9
  Day 21: Missing | 52 | 57
  Day 28: 0 = No clinical or virological evidence of infection | 123 | 134
  Day 28: 1 = No limitations of activities | 23 | 13
  Day 28: 2 = Limitation of activities | 85 | 95
  Day 28: 3 = Hospitalised - no oxygen therapy | 0 | 0
  Day 28: 4 = Oxygen by mask, or nasal prongs | 3 | 2
  Day 28: 5 = Non-invasive ventilation, or high flow oxygen | 4 | 0
  Day 28: 6 = Intubation and mechanical ventilation | 0 | 1
  Day 28: 7 = Ventilation plus additional organ support | 1 | 3
  Day 28: 8 = Death | 14 | 14
  Day 28: Missing | 56 | 52
  Day 35: 0 = No clinical or virological evidence of infection | 147 | 153
  Day 35: 1 = No limitations of activities | 10 | 16
  Day 35: 2 = Limitation of activities | 71 | 73
  Day 35: 3 = Hospitalised - no oxygen therapy | 0 | 0
  Day 35: 4 = Oxygen by mask, or nasal prongs | 2 | 1
  Day 35: 5 = Non-invasive ventilation, or high flow oxygen | 1 | 0
  Day 35: 6 = Intubation and mechanical ventilation | 2 | 1
  Day 35: 7 = Ventilation plus additional organ support | 1 | 1
  Day 35: 8 = Death | 14 | 17
  Day 35: Missing | 61 | 52

9. Secondary Outcome: Change From Baseline in Total Score According to the Breathlessness, Cough and Sputum Scale (BCSS)
Description: The efficacy of SNG001 compared with placebo in patients with moderate COVID-19 by assessing changes in daily breathlessness, cough and sputum scores on a scale of 0 (no symptoms) up to 4 (severe symptoms) was evaluated. Breathlessness, Cough and Sputum is graded on a score from 0 to 4, where a higher score indicates worse symptoms. The total score is calculated by summing the individual scores and is therefore graded on a scale from 0 to 12.
  Change in value of BCSS total scale, with negative value indicates an improvement in symptoms.
Time Frame: Baseline to Day 15
Population: The ITT analysis population consisted of all randomised patients.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 309 | 314
score on a scale | -2.1 (0.09) | -2.2 (0.09)
Statistical Analysis 1: Comparison: SNG001 vs Placebo; SNG001 vs Placebo; Test type: Other; p = 0.410, Mixed Models Analysis; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.1 to 0.3], Standard Error of Mean 0.12

10. Secondary Outcome: Change From Baseline in National Early Warning Score (NEWS2) During the Hospitalisation Period
Description: The efficacy of SNG001 compared to placebo in patients with moderate COVID-19 by assessing changes in NEWS2 during hospitalisation period was evaluated. It is the sum of scores calculated for Respiratory rate, Oxygen Saturation, Systolic BP, Pulse and Temperature when graded on a scale from 0 to 3 where 0 means a normal assessment and a higher score indicates a greater deviation from normal . 2 more points are added if the patient is receiving oxygen and 3 further points are added if the patient has new-onset confusion, disorientation and/or agitation, where previously their mental state was normal. This gives a score between 0 and 20. Higher scores indicates high clinical risk.
  Change from baseline in NEWS-2 score, in negative values favors improvement.
Time Frame: Day 1 until Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 75 | 87
score on a scale
  Day 7 | -0.7 (3.08) | -0.7 (2.55)
  Day 14: number analyzed (Participants) | 17 | 30
  Day 14 | 0.2 (3.83) | -0.3 (3.32)
  Day 21: number analyzed (Participants) | 10 | 12
  Day 21 | 2.8 (3.16) | 2.3 (3.62)
  Day 28: number analyzed (Participants) | 4 | 6
  Day 28 | -0.5 (2.08) | 4.5 (4.37)

11. Secondary Outcome: Number of Patients With Presence of COVID-19 Symptoms Based on Daily Assessment
Description: The efficacy of SNG001 compared to placebo in patients with moderate COVID-19 by daily assessment of COVID-19 symptoms was evaluated. The presence of COVID-19 symptoms were assessed. Individual symptoms related to COVID-19/SARS-CoV-2 infection such as fever, breathlessness, and fatigue were assessed.
Time Frame: Day 1 until Day 90
Population: The ITT analysis population consisted of all randomised patients.
Measure: Count of Participants; unit: Participants
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 309 | 314
Participants
  Baseline | 306 | 310
  Day 7: number analyzed (Participants) | 264 | 271
  Day 7 | 221 | 234
  Day 14: number analyzed (Participants) | 247 | 251
  Day 14 | 169 | 162
  Day 21: number analyzed (Participants) | 243 | 238
  Day 21 | 154 | 139
  Day 28: number analyzed (Participants) | 236 | 243
  Day 28 | 122 | 117
  Day 35: number analyzed (Participants) | 164 | 171
  Day 35 | 61 | 69
  Day 60: number analyzed (Participants) | 166 | 171
  Day 60 | 44 | 57
  Day 90: number analyzed (Participants) | 176 | 176
  Day 90 | 41 | 51

12. Secondary Outcome: Number of Patients With Limitations of Usual Activities Based on Daily Assessment
Description: The efficacy of SNG001 compared to placebo in patients with moderate COVID-19 by daily assessment of limitation of usual activities was evaluated. The patients with limitations of usual activities were the patients who were unable to do usual activities (work, study, housework, family or leisure activities).
Time Frame: Day 1 until Day 35
Population: The ITT analysis population consisted of all randomised patients.
Measure: Count of Participants; unit: Participants
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 309 | 314
Participants
  Day 1 | 0 | 1
  Day 7: number analyzed (Participants) | 275 | 282
  Day 7 | 115 | 114
  Day 14: number analyzed (Participants) | 262 | 268
  Day 14 | 135 | 127
  Day 21: number analyzed (Participants) | 257 | 257
  Day 21 | 109 | 114
  Day 28: number analyzed (Participants) | 253 | 262
  Day 28 | 85 | 95
  Day 35: number analyzed (Participants) | 248 | 262
  Day 35 | 71 | 73

13. Secondary Outcome: Quality of Life Measured Using EuroQol 5-dimension 5-level (EQ-5D-5L)
Description: The efficacy of SNG001 compared to placebo in patients with moderate COVID-19 by using EQ-5D-5L was evaluated. The EQ-5D-5L provides a simple descriptive profile and a single index value for health status. The EQ-5D-5L self-rated questionnaire includes a visual analogue scale, which records the respondent's self-rated health status on a graduated (0-100) scale, with higher scores for higher health-related quality of life. It also includes the EQ-5D-5L descriptive system, which comprises 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The responses record five levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension. Here, 100 means the best health and 0 means the worst health.
Time Frame: Day 0, Day 7, Day 15, Day 28, Day 60 and Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 302 | 311
score on a scale
  Day 0 | 56.4 (21.72) | 56.9 (20.95)
  Day 7: number analyzed (Participants) | 259 | 264
  Day 7 | 72.6 (18.39) | 71.1 (20.44)
  Day 15: number analyzed (Participants) | 241 | 251
  Day 15 | 79.5 (18.25) | 79.0 (16.51)
  Day 28: number analyzed (Participants) | 234 | 242
  Day 28 | 83.3 (16.00) | 83.5 (14.90)
  Day 60: number analyzed (Participants) | 230 | 232
  Day 60 | 88.9 (14.16) | 88.0 (13.56)
  Day 90: number analyzed (Participants) | 233 | 229
  Day 90 | 90.3 (12.65) | 89.9 (13.65)

14. Secondary Outcome: General Anxiety Disorder 7 Questionnaire (GAD-7) Total Score
Description: The efficacy of SNG001 compared to placebo in patients with moderate COVID-19 by assessing long-COVID-19 symptoms was evaluated. Assessment of long-COVID-19 symptoms based on GAD-7 scale. GAD-7 scores seven individual item scales by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all", "several days", "more than half the days", and "nearly every day", respectively. The GAD-7 total score is calculated by summing the individual item scales to give a total score between 0 and 21. Higher score indicates severe anxiety.
Time Frame: Day 15, Day 28, Day 60 and Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 238 | 249
score on a scale
  Day 15 | 3.3 (4.08) | 3.5 (4.30)
  Day 28: number analyzed (Participants) | 231 | 240
  Day 28 | 2.2 (3.67) | 1.9 (3.29)
  Day 60: number analyzed (Participants) | 229 | 231
  Day 60 | 1.4 (3.06) | 1.7 (3.38)
  Day 90: number analyzed (Participants) | 228 | 227
  Day 90 | 1.0 (2.41) | 1.6 (3.43)

15. Secondary Outcome: Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-FS [Version 4]) Total Score
Description: Long-COVID-19 symptoms based on FACIT Fatigue Scale (Version 4) were evaluated. The FACIT Fatigue Scale (Version 4) included statements for patients such as: I feel fatigued; I feel weak all over; I feel listless ("washed out"); I feel tired; I have trouble starting things because I am tired; I have trouble finishing things because I am tired; I have energy; I am able to do my usual activities; I need to sleep during the day; I am too tired to eat; I need help doing my usual activities; and I am frustrated by being too tired to do the things I want to do. Based on responses on above statements, scoring was done and scores ranges from 0 to 4, where 0 represents not at all bothered by any of the above problems and 4 indicates very much bothered every day by any of the above problems. Total scores will be calculated as per the algorithm to give a total score on a scale between 0 and 52, where a higher total score indicates lower level of fatigue.
Time Frame: Day 15, Day 28, Day 60 and Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 239 | 248
score on a scale
  Day 15 | 39.1 (9.79) | 38.7 (10.31)
  Day 28: number analyzed (Participants) | 233 | 237
  Day 28 | 42.5 (10.19) | 42.8 (8.98)
  Day 60: number analyzed (Participants) | 228 | 230
  Day 60 | 46.4 (8.22) | 45.5 (7.96)
  Day 90: number analyzed (Participants) | 230 | 229
  Day 90 | 46.9 (8.01) | 46.3 (7.78)

16. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9) Total Score
Description: Long-COVID-19 symptoms based on PHQ-9 were evaluated. Patient Health Questionnaire-9 (PHQ-9) scores nine individual item scales by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all", "several days", "more than half the days", and "nearly every day", respectively. PHQ-9 total scores are calculated by summing the individual item scales to give a total score between 0 and 27. Higher scores indicated worse outcome.
Time Frame: Day 15, Day 28, Day 60 and Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 237 | 245
score on a scale
  Day 15 | 4.6 (4.47) | 5.0 (4.71)
  Day 28: number analyzed (Participants) | 232 | 238
  Day 28 | 3.2 (4.15) | 3.1 (4.02)
  Day 60: number analyzed (Participants) | 228 | 229
  Day 60 | 1.7 (3.23) | 2.1 (3.85)
  Day 90: number analyzed (Participants) | 229 | 228
  Day 90 | 1.5 (3.05) | 2.0 (3.89)

17. Secondary Outcome: Overall Pain Severity as Measured by Brief Pain Inventory Composite Scores
Description: Brief Pain Inventory Composite Scores is a self administered questionnaire that assesses pain interference. Overall pain severity score is calculated as the mean of questions of the brief pain inventory. The overall pain severity score is the average pain, on a scale from 0 to 10 of the worst pain, least pain and average pain in the last 24 hours and pain right now scores. Here, 0 indicates "No pain" and 10 indicates "Worst pain".
Time Frame: Day 15, Day 28, Day 60 and Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 50 | 55
score on a scale
  Day 15 | 3.4 (2.13) | 3.3 (1.98)
  Day 28: number analyzed (Participants) | 34 | 38
  Day 28 | 3.2 (1.98) | 3.2 (1.77)
  Day 60: number analyzed (Participants) | 21 | 20
  Day 60 | 4.1 (1.54) | 3.3 (1.94)
  Day 90: number analyzed (Participants) | 21 | 21
  Day 90 | 4.5 (2.14) | 3.5 (2.33)

18. Secondary Outcome: Number of Patients With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: The general safety and tolerability of SNG001 compared to placebo when administered to patients with moderate COVID-19 by assessing number of patients with AEs was assessed.
Time Frame: From the day informed consent is obtained until 28 days after the last administration of the study medication (Day 90)
Population: The Safety analysis population included all patients in the ITT population who receive at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SNG001 | Placebo
Number analyzed (Participants) | 301 | 303
Participants
  Any Treatment-emergent adverse event (TEAE) | 251 | 251
  Any serious TEAE | 38 | 55
  Any serious related TEAE | 3 | 3
  Any fatal TEAE | 16 | 16
  Any fatal TEAE related to study treatment | 0 | 0
  Any TEAE related to study treatment | 68 | 77
  Any TEAE leading to discontinuation of study treatment | 24 | 23
  Any Adverse Events of Note | 0 | 1

ADVERSE EVENTS:
Time Frame: From the day informed consent is obtained until 28 days after the last administration of the study medication (Day 90).
Description: For All Cause Mortality, ITT population was used which consisted of all the randomised patients.
  There were two patients randomised to placebo, one of which was never dosed and the other was dosed but the fatal Adverse Event (AE) started before dosing (i.e. not treatment emergent).
  For adverse event reporting (serious AEs and other AEs), safety analysis population was used.
  Safety analysis population included all patients in the ITT population who received at least one dose of the study drug.
Groups:
- SNG001: Patients received SNG001 via inhalation using Ultra nebuliser, once a day for 14 days
- Placebo: Patients received Placebo via inhalation using Ultra nebuliser, once a day for 14 days
Arm/Group | SNG001 | Placebo
All-Cause Mortality (participants affected / at risk) | 16/309 | 18/314
Serious Adverse Events (participants affected / at risk) | 38/301 | 55/303
Other Adverse Events (participants affected / at risk) | 250/301 | 248/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SNG001 (N=301) | Placebo (N=303)
COVID-19 (Infections and infestations) | 11 (11) | 8 (8)
COVID-19 pneumonia (Infections and infestations) | 8 (8) | 8 (8)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia acinetobacter (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (9)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
Oxygen consumption increased (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SNG001 (N=301) | Placebo (N=303)
Headache (Nervous system disorders) | 71 (84) | 61 (76)
Anosmia (Nervous system disorders) | 18 (18) | 20 (20)
Ageusia (Nervous system disorders) | 13 (13) | 18 (19)
Ear pain (Ear and labyrinth disorders) | 25 (26) | 9 (9)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 70 (78) | 72 (85)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 58 (62) | 54 (55)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 55 (57) | 47 (50)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 45 (54) | 35 (45)
Cough (Respiratory, thoracic and mediastinal disorders) | 39 (46) | 28 (32)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 (35) | 41 (46)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 22 (22)
Diarrhoea (Gastrointestinal disorders) | 22 (23) | 26 (31)
Constipation (Gastrointestinal disorders) | 21 (23) | 22 (27)
Vomiting (Gastrointestinal disorders) | 21 (22) | 23 (26)
Myalgia (Musculoskeletal and connective tissue disorders) | 60 (62) | 60 (65)
Arthralgia (Musculoskeletal and connective tissue disorders) | 54 (62) | 54 (62)
Fatigue (General disorders) | 39 (40) | 40 (43)
Chest pain (General disorders) | 36 (37) | 52 (54)
Pyrexia (General disorders) | 23 (25) | 30 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document is the property of Synairgen Research Ltd and may not be used, divulged, published, or otherwise disclosed with.

DOCUMENTS (2):
  • Study Protocol (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT04732949/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT04732949/SAP_001.pdf